CLINICAL TRIAL: NCT07237139
Title: Intrapulmonary Volume Changes During Synchronized Noninvasive Positive Pressure Ventilation In Preterm Infants
Brief Title: Pulmonary Volume Changes During Synchonized Noninvasive Positive Pressure Ventilation
Acronym: INSPIRE
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: University Hospital, Zürich (Other)
Responsible Party: Sponsor
Other Study IDs: INSPIRE
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Infant, Preterm; Respiratory Distress Syndrome (Neonatal); Chronic Lung Disease of Newborn; Respiratory Support; Synchronized Noninvasive Positive Pressure Ventilation (SNIPPV); Lung Volume
Keywords: Synchronized noninvasive positive pressure ventilation (SNIPPV); Lung volume; Electrical Impedance Tomography (EIT); infant, preterm
MeSH Terms: conditions — Premature Birth; Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preterm infants with a gestational age < 30 0/7 weeks at birth: Infants on sNIPPV respiratory support and below 4 weeks chronological age
  Interventions: Device: Electrical Impedance Tomography (EIT)

INTERVENTIONS:
Device: Electrical Impedance Tomography (EIT) — Electrical Impedance Tomography and clinical data will be recorded continuously. Corresponding data will be extracted and analyzed at five pre-defined timepoints.

SUMMARY:
Current evidence suggests that noninvasive positive pressure ventilation (NIPPV) is more effective than continuous positive airway pressure (CPAP) in preventing respiratory failure in preterm infants with respiratory distress syndrome (RDS), both as initial and post-extubation support. NIPPV may be delivered in synchronized (sNIPPV) or non-synchronized (nsNIPPV) modes, with sNIPPV offering clear benefits by coordinating support with the infant's own breathing. Recent studies indicate sNIPPV is superior to nsNIPPV in preventing respiratory failure, though the intrapulmonary mechanisms behind this advantage remain unclear. To address this, the present study uses Electrical Impedance Tomography (EIT) to evaluate how lung volume changes during different types of breaths and ventilator inflations - spontaneous breaths, synchronized inflations, non-synchronized inflations, and backup inflations - in preterm infants receiving sNIPPV.

DETAILED DESCRIPTION:
Hypothesis:

Synchronized inflations during NIPPV will increase tidal volumes (VT) and lung aeration when compared with non-synchronized inflations. Pressure peaks delivered during expiration (non-synchronized inflations), between spontaneous breaths (backup inflations), or during periods of apnea (backup inflations) will not increase relative VT.

Primary objective:

The primary objective is to assess lung volume changes between spontaneous breaths and synchronized inflations, non-synchronized inflations, and backup inflations using EIT.

Secondary objectives:

The secondary objectives are to assess regional differences in aeration and ventilation among spontaneous breaths, synchronized inflations, non-synchronized inflations, and backup inflations using EIT.

Primary endpoint:

Difference in relative Vt (rel. Delta-Z) between spontaneous breaths and synchronized inflations.

Study procedures:

Study procedures include attaching an EIT belt and a pulse oximeter sensor during the final nursing care session before the study begins. Synchronized NIPPV is provided by EVEneo ventilators, and synchronization will be achieved through an abdominal capsule (Graseby).

1. Sixty minutes after the beginning of the EIT recording , the noninvasve ventilation mode will be switched to CPAP for 2 minutes. This 2-minute period will be the baseline period during which spontaneous breathing will be assessed.
2. The NIV mode will then be switched back to sNIPPV. Ventilator settings will be maintained at the same levels used before the start of the study, and adjustments will not be permitted.
3. Prior to the next nursing care session, a second 2-minute nCPAP period will be introduced and serve as the baseline (together with the 1st CPAP period) .
4. The EIT recording and SpO2/HR measurements will continue until the next nursing care round, at which point the EIT belt and SpO2 sensor will be removed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent by one or both parents or legal guardians
* Gestational age at birth < 30 0/7 weeks
* Infants on sNIPPV respiratory support
* Below 4 weeks chronological age

Exclusion Criteria:

* Severe congenital malformation adversely affecting lung aeration or perfusion (e.g., congenital heart defects)
* Too ill/unstable in the opinion of the treating physician.

Max Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will take place at the Department of Neonatology of the University Hospital Zurich. Preterm infants on a synchronized mode of non-invasive positive pressure ventilation will be screened for eligibility and parents will be approached by the treating physician or a clinician-researcher who is authorized to access the patient's clinical data.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Tidal volume (VT) | At five pre-defined timepoints from the beginning to the end of the study at 180 minutes.
  Difference in relative VT (rel. ΔZ) between spontaneous breaths and synchronized inflations.

SECONDARY OUTCOMES:
Global lung impedance | At five pre-defined timepoints from the beginning to the end of the study at 180 minutes.
  Difference between end-expiratory lung impedance (EELI) and inspiratory onset lung impedance (SILI) during spontaneous breaths, synchronized inflations, non-synchronized inflations, and back-up inflations.
Regional tidal volume distribution | At five pre-defined timepoints from the beginning to the end of the study at 180 minutes.
  Difference in regional tidal distribution between spontaneous breaths, synchronized inflations, non-synchronized inflations and back-up inflations
Center of ventilation | At five pre-defined timepoints from the beginning to the end of the study at 180 minutes.
  Difference in center of ventilation between spontaneous breaths, synchronized inflations, non-synchronized inflations and back-up inflations
Silent spaces | At five pre-defined timepoints from the beginning to the end of the study at 180 minutes.
  Difference in silent spaces between spontaneous breaths, synchronized inflations, non-synchronized inflations and back-up inflations
Global inhomogeneity index | At five pre-defined timepoints from the beginning to the end of the study at 180 minutes.
  Difference in global inhomogeneity index between spontaneous breaths, synchronized inflations, non-synchronized inflations and back-up inflations. An inhomogeneity index of zero represents a perfectly homogeneous distribution of ventilation.
Coefficient of variation | At five pre-defined timepoints from the beginning to the end of the study at 180 minutes.
  Difference in coefficient of variation (EIT) between spontaneous breaths, synchronized inflations, non-synchronized inflations and back-up inflations
Inspiratory time | At five pre-defined timepoints from the beginning to the end of the study at 180 minutes.
  Difference in inspiratory times between spontaneous breaths, synchronized inflations, non-synchronized inflations and back-up inflations
Expiratory time | At five pre-defined timepoints from the beginning to the end of the study at 180 minutes.
  Difference in expiratory times between spontaneous breaths, synchronized inflations, non-synchronized inflations and back-up inflations
Lung ultrasound score | Immediately before the first infant handling as well as following electrical impedance tomography belt removal.
  Difference in lung ultrasound score at two pre-defined timepoints.
  Each lung will be divided into 3 areas. For each lung area, a 0- to 3-point score will be given (total score ranging from 0-18). Higher scores represent greater severity of lung disease.
Heart rate | Continuous measurement during the 180-minute recording period.
  Changes of heart rate between five pre-defined time points.
Peripheral oxygen saturation | Continuous measurement during the 180-minute recording period.
  Changes in oxygen saturation between five pre-defined time points.
Oxygen supplementation | Continuous measurement during the 180-minute recording period.
  Changes in FiO2 between five pre-defined time points.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Cannizzaro, MD, Study Chair — Newborn Research, Department of Neonatology, University Hospital and University of Zurich, Zurich, Switzerland
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No